CLINICAL TRIAL: NCT03381742
Title: Efficacy and Safety of Different Ticagrelor Regimens Versus Clopidogrel in Patients With Coronary Artery Disease: a Retrospective Multicenter Study (SUPERIOR)
Brief Title: Efficacy and Safety of Low-dose Ticagrelor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Central Hospital of Jia Mu Si City (Unknown); First Affiliated Hospital of Kunming Medical University (Other); RenJi Hospital (Other); Tianjin Medical University General Hospital (Other); Weifang People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shengjing Hospital (Other); Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACS-2
Record Dates: First submitted 2017-12-14; First posted 2017-12-22 (Actual); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ticagrelor 45mg bidpo. (Experimental): To observe the efficacy and safety of ticagrelor 45mg bidpo. in patients with coronary artery disease.
  Interventions: Drug: Ticagrelor
- ticagrelor 90mg qdpo. (Experimental): To observe the efficacy and safety of ticagrelor 90mg qdpo. in patients with coronary artery disease.
  Interventions: Drug: ticagrelor
- ticagrelor 90mg bidpo. (Active Comparator): To observe the efficacy and safety of ticagrelor 90mg bidpo. in patients with coronary artery disease.
  Interventions: Drug: ticagrelor
- clopidogrel 75mg qdpo. (Active Comparator): To observe the efficacy and safety of clopidogrel 75mg qdpo. in patients with coronary artery disease.
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — ticagrelor 45 mg twice daily for 5 consecutive days at least.
  Arms: ticagrelor 45mg bidpo.
Drug: ticagrelor — ticagrelor 90 mg once daily for 5 consecutive days at least.
  Arms: ticagrelor 90mg qdpo.
Drug: ticagrelor — ticagrelor 90 mg twice daily for 5 consecutive days at least.
  Arms: ticagrelor 90mg bidpo.
Drug: clopidogrel — clopidogrel 75 mg once daily for 5 consecutive days at least.
  Arms: clopidogrel 75mg qdpo.

SUMMARY:
Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. Recent study found that ticagrelor 90mg twice a day orally could significantly reduce the occurrence of clopidogrel resistance and adverse cardiovascular events. The previous studies have reported that half-dose ticagrelor had the similar inhibitory effect on platelet aggregation as the standard-dose ticagrelor, which was significantly stronger than that in the clopidogrel group. One-quarter standard-dose ticagrelor provided greater degree of platelet inhibition than standard dose clopidogrel in Chinese patients with stable CAD. But large-scale clinical trials are still needed to confirm the effects of low-dose ticagrelor on platelet function in Chinese patients with coronary heart disease.

DETAILED DESCRIPTION:
Dual Antiplatelet Therapy (DAPT) with aspirin and P2Y12 receptor inhibitor remains a cornerstone in the secondary prevention of coronary artery disease (CAD). Clopidogrel is one of the most commonly used antithrombotic agent that inhibits the platelet P2Y(12) adenosine diphosphate (ADP) receptor.

Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. Recent study found that ticagrelor 90mg twice a day orally could significantly reduce the occurrence of clopidogrel resistance and adverse cardiovascular events. The previous studies have reported that half-dose ticagrelor had the similar inhibitory effect on platelet aggregation as the standard-dose ticagrelor, which was significantly stronger than that in the clopidogrel group. One-quarter standard-dose ticagrelor provided greater degree of platelet inhibition than standard dose clopidogrel in Chinese patients with stable CAD. But large-scale clinical trials are still needed to confirm the effects of low-dose ticagrelor on platelet function in Chinese patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease

Exclusion Criteria:

* younger than 18 years of age;
* anti-platelet therapy with clopidogrel or ticagrelor for less than 5 days;
* previous or current treatment with any other potentially confounding drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3043 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, MD, Principal Investigator — Cardiovascular Department, the First Affiliated Hospital of Harbin Medical University
Locations (1):
- Thromboela-Stogram, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3,737 CAD patients who received either clopidogrel or ticagrelor therapy and underwent TEG test from 11 medical centers. Among these patients, 1,725 subjects were treated with clopidogrel and 2,012 subjects were treated with different ticagrelor regimens.
Period: Overall Study
Arm/Group | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Bidpo. | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Qdpo.
Started | 525 | 501 | 1511 | 506
Completed | 525 | 501 | 1511 | 506
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo. | Total
Number analyzed (Participants) | 1511 | 501 | 525 | 506 | 3043
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [55 to 69] | 61 [52 to 67] | 62 [55 to 69] | 62 [55 to 68] | 62 [55 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 159 | 201 | 237 | 1129
  Male | 979 | 342 | 324 | 269 | 1914
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1511 | 501 | 525 | 506 | 3043
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 1511 | 501 | 525 | 506 | 3043
Weight [Median (Inter-Quartile Range); unit: kg] | 70 [63 to 78] | 70 [62 to 78] | 70 [60 to 75] | 70 [60 to 75] | 70 [62 to 78]
smoking [Count of Participants; unit: Participants] | 736 | 234 | 226 | 202 | 1398
Hypertension [Count of Participants; unit: Participants] | 879 | 243 | 332 | 287 | 1741
diabetes mellitus [Count of Participants; unit: Participants] | 426 | 126 | 161 | 117 | 830
chronic kidney disease [Count of Participants; unit: Participants] | 60 | 13 | 25 | 13 | 111
percutaneous coronary intervention [Count of Participants; unit: Participants] | 1056 | 326 | 241 | 179 | 1802
coronary artery bypass grafting [Count of Participants; unit: Participants] | 12 | 2 | 2 | 1 | 17
total cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 4.2 [3.4 to 5.1] | 3.9 [2.6 to 5] | 4.3 [3.4 to 5.3] | 4.7 [3.8 to 5.7] | 4.24 [3.39 to 5.18]
triglyceride [Median (Inter-Quartile Range); unit: mmol/L] | 1.6 [1.2 to 2.4] | 1.9 [1.3 to 3.6] | 1.7 [1.2 to 2.7] | 1.6 [1.1 to 2.4] | 1.67 [1.17 to 2.57]
high density lipoprotein [Median (Inter-Quartile Range); unit: mmol/L] | 1.1 [0.9 to 1.3] | 1.1 [0.9 to 1.3] | 1.1 [1.0 to 1.3] | 1.2 [1 to 1.4] | 1.1 [0.93 to 1.3]
low density lipoprotein [Median (Inter-Quartile Range); unit: mmol/L] | 2.6 [2.1 to 3.2] | 2.8 [2.1 to 3.3] | 2.7 [2.2 to 3.3] | 2.9 [2.4 to 3.6] | 2.68 [2.17 to 3.25]
creatinine [Median (Inter-Quartile Range); unit: μmol/L] | 71 [61.4 to 82.9] | 69.7 [59.2 to 81] | 68.7 [59.1 to 80.7] | 67.7 [57.6 to 79.6] | 69.9 [59.5 to 81.7]
uric acid [Median (Inter-Quartile Range); unit: μmol/L] | 330 [276 to 390] | 338 [280 to 408] | 323 [268 to 385] | 320 [266 to 387] | 328.4 [271.5 to 391.8]
aspirin use [Count of Participants; unit: Participants] | 1429 | 446 | 475 | 443 | 2793
acute myocardial infarction [Count of Participants; unit: Participants] | 568 | 180 | 98 | 49 | 895

OUTCOME MEASURES:

1. Primary Outcome: ADP-induced Inhibition of Platelet Aggregation
Description: The venous blood samples for platelet function test were drawn after an overnight fast, at 12 hours post-last study-drug dose for subjects receiving twice-daily administrations, and at 24 hours post-last study-drug dose for subjects treated with once-daily regimens. The blood was collected in an evacuated vacuum tube containing 3.2% trisodium citrate and lithium heparin. Then the samples were processed within two hours of blood draw according to standard operating procedure. The physical properties of samples were analyzed using Thromboelastography (TEG) Hemostasis Analyzer (CFMS LEPU-8800, Lepu Medical Technology Co., Ltd, Beijing, China) and automated analytical software. TEG test used four channels to detect the effects of anti-platelet therapy via the arachidonic acid (AA) and ADP pathways. TEG test results were expressed in terms of ADP-induced inhibition of platelet aggregation (IPA, range 0% - 100%), with higher values indicating greater platelet inhibition.
Time Frame: up to 5 days
Measure: Median (Inter-Quartile Range); unit: percentage of inhibition of platelet agg
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
percentage of inhibition of platelet agg | 54.9 [31.9 to 79.1] | 80.6 [64.1 to 94] | 73.6 [52.6 to 93.7] | 66 [46.9 to 87]

2. Primary Outcome: Number of Participants With Bleeding (Major or Minor Bleeding)
Description: Major bleeding was defined as type ≥ 3 and minor bleeding as types 1 and 2, in accordance to the Bleeding Academic Research Consortium classification. (Mehran R et al. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449.)
Time Frame: up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
Participants
  Minor bleeding | 15 | 30 | 14 | 9
  Major bleeding | 0 | 0 | 0 | 0
  No bleeding | 1496 | 471 | 511 | 497

3. Secondary Outcome: ADP-induced Platelet-fibrin Clot Strength (MA)
Description: The physical properties of samples were analyzed using Thromboelastography (TEG) Hemostasis Analyzer (CFMS LEPU-8800, Lepu Medical Technology Co., Ltd, Beijing, China) and automated analytical software. TEG test used four channels to detect the effects of anti-platelet therapy via the arachidonic acid (AA) and ADP pathways. TEG test results were expressed in terms of ADP-induced platelet-fibrin clot strength (MA). A MA>47mm was shown to have a high predictive value for 3-year post-PCI ischemic events during dual antiplatelet therapy. Moreover, ROC curve and quartile analysis suggested MA<31 mm as a predictive value for post-PCI bleeding events (J Am Coll Cardiol. 2013;62(24):2261-73. doi: 10.1016/j.jacc.2013.07.101.).
Time Frame: up to 5 days
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
mm | 40.3 [27 to 51.6] | 28.4 [18.5 to 38.9] | 32.3 [19.5 to 43.9] | 34.05 [23.6 to 46.1]

4. Secondary Outcome: Number of Participants With High On-Treatment Platelet Reactivity (HTPR)
Description: HTPR was defined as IPA ≤ 30% and MA ≥ 47 mm.
Time Frame: up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
Participants
  HTPR | 317 | 13 | 23 | 32
  Non-HTPR | 1194 | 488 | 502 | 474

5. Secondary Outcome: Number of Participants With Cardiovascular Event (Cardiovascular Death, New-onset Myocardial Infarction, or Stroke)
Description: Cardiovascular death was defined as sudden cardiac death, fatal myocardial infarction, death due to heart failure, or death due to other cardiovascular causes. Stroke was defined as the focal loss of neurologic function caused by an ischemic or a hemorrhagic event with residual symptoms lasting at least 24 hours or eventually leading to death.
Time Frame: up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
Participants
  Participants with cardiovascular death | 0 | 0 | 0 | 0
  Participants without cardiovascular events | 1511 | 501 | 525 | 506
  Participants with new-onset myocardial infarction | 0 | 0 | 0 | 0
  Participants with stroke | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With New-onset Dyspnea
Description: New-onset dyspnea in patients without previous history of dyspnea
Time Frame: up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
Number analyzed (Participants) | 1511 | 501 | 525 | 506
Participants
  Participants with new-onset dyspnea | 34 | 29 | 32 | 28
  Participants without new-onset dyspne | 1477 | 472 | 493 | 478

ADVERSE EVENTS:
Time Frame: up to 5 days
Arm/Group | Clopidogrel 75mg Qdpo. | Ticagrelor 90mg Bidpo. | Ticagrelor 45mg Bidpo. | Ticagrelor 90mg Qdpo.
All-Cause Mortality (participants affected / at risk) | 0/1511 | 0/501 | 0/525 | 0/506
Serious Adverse Events (participants affected / at risk) | 0/1511 | 0/501 | 0/525 | 0/506
Other Adverse Events (participants affected / at risk) | 0/1511 | 0/501 | 0/525 | 0/506

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03381742/Prot_SAP_000.pdf